CLINICAL TRIAL: NCT03838276
Title: Ponderal Outcomes After Roux-en-Y Gastric Bypass With Alimentary Limb (AL) of 150cm and Biliopancreatic Limb (BPL) of 100cm vs AL 100cm and BPL 150cm
Brief Title: RYGB AL 150cm BPL 100cm vs RYGB AL 100cc BPL 150cm
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Department of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRJC 19-21
Record Dates: First submitted 2019-02-09; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AL150 BPL100 (Active Comparator): Roux-en-Y gastric bypass with 150cm of alimentary limb and 100cm of biliopancreatic limb
  Interventions: Procedure: AL 150 BPL100
- AL100 BPL150 (Experimental): Roux-en-Y gastric bypass with 100cm of alimentary limb and 150cm of biliopancreatic limb
  Interventions: Procedure: AL 100 BPL 150

INTERVENTIONS:
Procedure: AL 150 BPL100 — Roux-en-Y gastric bypass with 150cm of alimentary limb and 100cm of biliopancreatic limb
  Arms: AL150 BPL100
Procedure: AL 100 BPL 150 — Roux-en-Y gastric bypass with 100cm of alimentary limb and 150cm of biliopancreatic limb
  Arms: AL100 BPL150

SUMMARY:
A Roux-en-Y gastric bypass will be performed in all the cases. Patients will be randomized according the limb lengths:

* Group 1: Alimentary limb (AL) 150cm and biliopancreatic limb (BPL) 100cm
* Group 2: AL 100cm and BPL 150cm

Weight loss will be evaluated 1 year after surgery

DETAILED DESCRIPTION:
A Roux-en-Y gastric bypass will be performed in all the cases. Patients will be randomized according the limb lengths:

* Group 1: Alimentary limb 150cm and biliopancreatic limb 100cm
* Group 2: Alimentary limb 100cm and biliopancreatic limb 150cm

Weight loss will be evaluated 1 year after surgery

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40 Kg/m2
* BMI > 35 Kg/m2, associated with obesity-related comorbidities
* Patients undergoing Roux-en-Y gastric bypass as bariatric procedure

Exclusion Criteria:

* Patients undergoing Roux-en-Y gastric bypass as revisional procedure
* Patients lost to follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 1 year after surgery
  Weight loss will be assessed 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Santiago de Battista, Study Chair — Hospital La PLata